CLINICAL TRIAL: NCT03072017
Title: Monitored Breathing Awareness Therapy for Insomnia Disorder in Older Adults: Phase 1 Open Label Pilot
Brief Title: Monitored Breathing Awareness Therapy for Insomnia Disorder in Older Adults
Acronym: MBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Advanced Medical Electronics (Other)
Responsible Party: Principal Investigator, Nalaka Gooneratne, Associate Professor, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 816717
Record Dates: First submitted 2017-02-27; First posted 2017-03-07 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBAT (Experimental): Monitored breathing awareness therapy administered using a mobile device on a nightly basis during sleep onset.
  Interventions: Behavioral: MBAT

INTERVENTIONS:
Behavioral: MBAT — Breathing-based intervention

SUMMARY:
Insomnia can be a chronic problem that leads to significant daytime fatigue, stress and numerous negative health consequences including depression. Advanced Medical Electronics, in partnership with researchers are the University of Pennsylvania, propose developing an innovative, non-drug, low-risk, intervention that can be implemented on mobile devices for the treatment of insomnia.

DETAILED DESCRIPTION:
Open-label pilot study in 20 older adults with insomnia (sleep onset latency>30 minutes for at least 3 nights a week) with a two week intervention period.

ELIGIBILITY:
Inclusion Criteria:

1) Sleep onset latency > 30 min for at least 3 nights per week

Exclusion Criteria:

1. Unable to perform tests due to inability to communicate verbally/blindness, inability to write and read in English (the study questionnaires are in English and do not exist in validated form for other languages).
2. Cognitive impairment; cognitively impaired patients may not be able to comply with the protocol).
3. History of a diagnosed non-insomnia sleep disorder, such as sleep apnea or circadian rhythm disorder
4. Upper extremity motor impairment that would preclude MBAT therapy (e.g., quadriplegia).

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Sleep onset latency | two weeks
  Time to fall asleep

IPD SHARING:
Plan to Share IPD: Yes
At conclusion of study as per NIH guidelines